CLINICAL TRIAL: NCT06681688
Title: Prospective Study of Complication Rates in Cataract Surgery Patients Treated With Combined Pre-operative NSAID, OMIDRIA, and Subconjunctival Triamcinolone Acetonide Compared With Peri-operative Standard of Care
Brief Title: Study of Complication Rates in Cataract Surgery Patients Treated With Combined Pre-operative NSAID, OMIDRIA, and Subconjunctival Triamcinolone Acetonide Compared With Peri-operative SOC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inder Paul Singh, M.D. (Other)
Collaborators: The Eye Associates (Other)
Responsible Party: Sponsor-Investigator, Inder Paul Singh, M.D., Principal Investigator, The Eye Centers of Racine and Kenosha
Organization: The Eye Centers of Racine and Kenosha (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSS V2 6324
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Cataract
Keywords: OMIDRIA
MeSH Terms: conditions — Cataract | interventions — Triamcinolone Acetonide; Phenylephrine; Ketorolac; Ketorolac Tromethamine; Moxifloxacin; prednisolone acetate; Drugs, Generic; Methylprednisolone

STUDY DESIGN:
Intervention Model Description: This is a 2-arm non-inferiority trial with the following arms:
  * Control arm: Participants undergoing cataract surgery using conventional standard of care peri-operative eyedrops.
  * Study arm: Participants undergoing cataract surgery with a regimen of peri-operative topical eyedrops administered to the participant by study staff, in combination with intracameral phenylephrine 1.0%/ketorolac 0.3%, subconjunctival triamcinolone acetonide, and intracameral moxifloxacin.
Who Masked: Investigator
Masking Description: The biostatistician analyzing the data will be masked to both treatment arm and surgery center.
  When the Investigators or Sponsor look at the data, they will also be masked to treatment arm and surgery center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Arm (OMIDRIA) (Experimental): * Pre-op, 1 drop ketorolac (0.5%) {Toradol}, 1 drop moxifloxacin (0.5%) {Avelox}
  * Prior to surgery: 1 drop ketorolac (0.5%), 1 drop moxifloxacin (0.5%)
  * Concl. of surgery while still in the OR: 1 drop ketorolac (0.5%), 1 drop moxifloxacin (0.5%), 1 drop prednisolone acetate (1%) {Pred Forte}
  * Post-op recovery: 1 drop ketorolac (0.5%), 1 drop moxifloxacin (0.5%), 1 drop prednisolone acetate (1%).
  Intraoperative interventions: intracameral phenylephrine {Sudafed} 1.0%/ketorolac 0.3%, {OMIDRIA} intracameral moxifloxacin (0.5%), and subconjunctival triamcinolone acetonide (0.4 mL, 10 mg/mL) {Kenalog}.
  In-office drops administered by study staff at the end of the 1-day visit: 1 drop ketorolac (0.5%), 1 drop moxifloxacin (0.5%), 1 drop prednisolone acetate (1%).
  Rescue therapy will be allowed, if necessary, at the discretion of the evaluating physician and will consist of prednisolone acetate (1%) QID (taper also at the discretion of the evaluating physician).
  Interventions: Drug: Omidria, {0.3%-1% Intraocular Solution}, VIGAMOX {0.5% moxifloxacin hydrochloride}, Kenalog {0.4 ml, 10mg/ml, triamcinolone acetonide}
- Control Arm (Standard of Care) (Active Comparator): Self-administration of:
  Ketorolac (0.5%) {Toradol} four times daily (QID) x 1 day and moxifloxacin (0.5%) {Avelox} drops three times daily (TID) x 1 day before SX.
  On the Day of SX, eyes will receive in-office drops administered by study staff according to the following:
  * In pre-operative holding: 1 drop ketorolac (0.5%), 1 drop moxifloxacin (0.5%)
  * Immediately prior to SX: 1 drop ketorolac (0.5%), 1 drop moxifloxacin (0.5%)
  * At the conclusion of SX while still in the operating room: 1 drop ketorolac (0.5%), 1 drop moxifloxacin (0.5%), 1 drop prednisolone acetate (1%) Pred Forte}
  * Any time in post-op recovery: 1 drop ketorolac (0.5%), 1 drop moxifloxacin (0.5%), 1 drop prednisolone acetate (1%).
  Eyes will then self-administer the following postoperative interventions: ketorolac drops QID x 1 month. Prednisolone acetate tapering QID x1 week, TID x 1 week, twice daily (BID) x 1 week, and once daily (QD) x 1 week; and moxifloxacin drops TID x 1 week.
  Interventions: Drug: Ketorolac (0.5%) {Toradol}, moxifloxacin (0.5%) {VIGAMOX}, prednisolone acetate (1%) {Pred Forte}

INTERVENTIONS:
Drug: Omidria, {0.3%-1% Intraocular Solution}, VIGAMOX {0.5% moxifloxacin hydrochloride}, Kenalog {0.4 ml, 10mg/ml, triamcinolone acetonide} — Eyes in the Study Arm will be treated with the following intraoperative interventions: Intracameral (OMIDRIA) phenylephrine 1.0%/ketorolac 0.3%, intracameral moxifloxacin (0.5%), and subconjunctival triamcinolone acetonide (0.4 mL, 10mgs/mL).
  Other Names: (OMIDRIA), Phenylephrine (1%) and Ketorolac (0.3%) intraocular solution
  Arms: Study Arm (OMIDRIA)
Drug: Ketorolac (0.5%) {Toradol}, moxifloxacin (0.5%) {VIGAMOX}, prednisolone acetate (1%) {Pred Forte} — On the Day of Surgery, eyes in the Control Arm will receive in-office drops administered by study staff according to the following schedule:
  * In pre-operative holding: 1 drop ketorolac (0.5%), 1 drop moxifloxacin (0.5%)
  * Immediately prior to surgery: 1 drop ketorolac (0.5%), 1 drop moxifloxacin (0.5%)
  * At the conclusion of surgery while still in the operating room: 1 drop ketorolac (0.5%), 1 drop moxifloxacin (0.5%), 1 drop prednisolone acetate (1%)
  * Any time in postoperative recovery: 1 drop ketorolac (0.5%), 1 drop moxifloxacin (0.5%), 1 drop prednisolone acetate (1%)
  Other Names: TORADOL (Generic), Vigamox, Avalox, Pred Forte, Prelone, Omnipred
  Arms: Control Arm (Standard of Care)

SUMMARY:
This is a multicenter, 2-arm, randomized, prospective study of patients slated for bilateral cataract extraction. One eye will be randomized to the Study Arm, and the fellow eye will be randomized to the Control Arm.

DETAILED DESCRIPTION:
For the control arm interventions:

Preoperatively, the Control Arm (control eye) will self-administer a regimen of ketorolac four times daily (QID) x 1 day and moxifloxacin drops three times daily (TID) x 1 day before surgery. On the Day of Surgery, eyes in the Control Arm will receive in-office drops administered by study staff according to the following schedule:

* In pre-operative holding: 1 drop ketorolac, 1 drop moxifloxacin
* Immediately prior to surgery: 1 drop ketorolac, 1 drop moxifloxacin
* At the conclusion of surgery while still in the operating room: 1 drop ketorolac, 1 drop moxifloxacin, 1 drop prednisolone acetate
* Any time in postoperative recovery: 1 drop ketorolac, 1 drop moxifloxacin, 1 drop prednisolone acetate

Eyes in the Control Arm will then self-administer the following postoperative interventions: ketorolac drops QID x 1 month, prednisolone acetate tapering QID x1 week, TID x 1 week, twice daily (BID) x 1 week, and once daily (QD) x 1 week; and moxifloxacin drops TID x 1 week.

For the study arm interventions:

Eyes will receive in-office drops on the Day of Surgery administered by study staff according to the following schedule:

* In pre-operative holding: 1 drop ketorolac, 1 drop moxifloxacin
* Immediately prior to surgery: 1 drop ketorolac, 1 drop moxifloxacin
* At the conclusion of surgery while still in the operating room: 1 drop ketorolac, 1 drop moxifloxacin, 1 drop prednisolone acetate
* Any time in postoperative recovery: 1 drop ketorolac, 1 drop moxifloxacin, 1 drop prednisolone acetate.

Eyes in the Study Arm will be treated with the following intraoperative interventions: intracameral phenylephrine 1.0%/ketorolac 0.3%, intracameral moxifloxacin, and subconjunctival triamcinolone acetonide.

The following study assessments will take place for all subjects:

Visual acuity measured by the Early Treatment of Diabetic Retinopathy Study (ETDRS) chart (pinhole visual acuity [VA] or best corrected visual acuity [BCVA])

* Slit lamp examination, including intraocular pressure (IOP) measurement
* Grading of inflammation
* Standard Patient Evaluation of Eye Dryness (SPEED) questionnaire
* Pain assessment on a 0-4 scale
* Overall participant satisfaction on a 0-10 scale
* Optical coherence tomography (OCT) imaging

Eyes in the Study Arm will also receive in-office drops administered by study staff at the end of the 1-day visit: 1 drop ketorolac, 1 drop moxifloxacin, 1 drop prednisolone acetate.

Rescue therapy for postoperative inflammation will be allowed for Study Arm participants, if necessary, at the discretion of the evaluating physician and will consist of prednisolone acetate QID (taper also at the discretion of the evaluating physician).

ELIGIBILITY:
Inclusion Criteria:

* Adult participants > 18 years of age undergoing bilateral cataract surgery
* Able to provide written informed consent prior to any study related procedure
* Able and willing, as assessed by the Investigator, to follow study instructions, complete study assessments, comply with the protocol, and attend study visits for the duration of the study
* Patients deemed to be "higher risk" for postoperative complications (e.g., well-controlled diabetes (HbA1c ≤7.0), history of uveitis, history of retinal vein occlusion, history of epiretinal membrane, history of vitreomacular traction, evidence of posterior synechiae, etc.) MAY be enrolled provided there has been no evidence of active disease or treatment in the prior 12 months
* Participants who do not meet the exclusion criteria may be enrolled.

Exclusion Criteria:

* Cataract surgery combined with any other procedure (e.g., glaucoma, retina, etc.)
* Glaucoma patients or known steroid responders
* Oral anti-inflammatory medications to treat a systemic disease (exceptions to this include 81 mg aspirin, ibuprofen for headache, etc.)
* Intraocular injection within 6 months
* Any prior ocular implant
* Diagnosis of retinal thickening in the study eye within 12 months of enrollment
* Inability to provide informed consent
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
inflammation | 8 days
  The proportion of participants with inflammation on Day 8. (Participants will be considered to have no inflammation (Grade 0) if they have ≤ 2 anterior chamber cells and are asymptomatic.) {Anterior Inflammation Scale, 0-4 with 4 being the worst or most severe score}

SECONDARY OUTCOMES:
SPEED Questionnaire | 30 days
  Mean change in SPEED Questionnaire from baseline to Day 8 and baseline to Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Paul Singh, MD, Principal Investigator — The Eye Centers of Racine & Kenosha
Locations (2):
- United States (2):
  - The Eye Associates - Venice, Venice, Florida
  - The Eye Centers of Racine & Kenosha, Racine, Wisconsin

IPD SHARING:
Plan to Share IPD: No